CLINICAL TRIAL: NCT04703595
Title: Chronic Cough and CANVAS (Cerebellar Ataxia With Neuropathy and Bilateral Vestibular Areflexia Syndrome): Screening for Mutations in Subunit 1 of the Replication Factor Complex: Initial Pilot Study
Brief Title: Chronic Cough and CANVAS (Cerebellar Ataxia With Neuropathy and Bilateral Vestibular Areflexia Syndrome)
Acronym: CANVAS
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TOS-2020-143
Record Dates: First submitted 2021-01-05; First posted 2021-01-11 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2022-07

CONDITIONS: Cough; Cerebellar Ataxia; Gastroesophageal Reflux
Keywords: Cerebellar Ataxia; chronic cough; CANVAS
MeSH Terms: conditions — Cough; Cerebellar Ataxia; Gastroesophageal Reflux; Chronic Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — For the molecular study of the DNA sample of the patients, two techniques will be used: amplification by standard Polymerase chain reaction with primers flanking the intron 2 fragment of the RFC1 gene and amplification by Repeated Primed Polymerase chain reaction in 3 independent reactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 50 non-smoking patients with chronic cough: 50 non-smoking patients aged between 30 and 99 years with chronic and / or refractory cough as the only manifestation or associated with gastroesophageal reflux
  Interventions: Genetic: To determine the presence of biallelic expansion of AAGGG in RFC1 in patients with chronic cough, regardless of the presence of neurological symptoms.

INTERVENTIONS:
Genetic: To determine the presence of biallelic expansion of AAGGG in RFC1 in patients with chronic cough, regardless of the presence of neurological symptoms. — To determine the presence of biallelic expansion of AAGGG in RFC1 in patients with chronic cough, regardless of the presence of neurological symptoms.
  For the molecular study of the DNA sample of the patients, two techniques will be used: standard Polymerase chain reaction amplification with primers flanking the intron 2 fragment of the RFC1 gene and amplification using Repeated Primed Polymerase chain reaction in 3 independent reactions.

SUMMARY:
Chronic cough is a frequent cause of Pneumology consultations. CANVAS syndrome (Cerebellar Ataxia with Neuropathy and bilateral Vestibular Areflexia Syndrome) is a progressive and disabling neurological disease that very frequently occurs with chronic cough. This cough invariably appears as a prodromal symptom that precedes neurological symptoms. The biallelic expansion of AAGGG in RFC1, a causal mutation in CANVAS syndrome, appears with high frequency in the general population. Objectives: Main: To determine the presence of biallelic expansion of AAGGG in RFC1 in patients with chronic cough, regardless of the presence of neurological symptoms. Secondary: Describe the phenotypic, functional and inflammatory characteristics of these patients. and Know the relationship between gastroesophageal reflux and chronic cough in patients with CANVAS. Method: A descriptive cross-sectional pilot study including 50 non-smoking patients between the ages of 30 and 99 years with chronic and / or refractory cough as the only manifestation or associated with gastroesophageal reflux. All patients will undergo the pertinent studies for the diagnosis of chronic cough, those who meet criteria for suspicion of gastroesophageal reflux will be requested an esophageal phmetry and esophageal manometry. Peripheral venous blood sample will be obtained for subsequent genetic analysis. Vibration sensitivity will be studied in all patients regardless of the presence of mutation. Those with alterations in vibratory sensitivity or mutations in RFC1 will be referred to the Neurology Service for a complementary neurological evaluation. For the molecular study of the DNA sample of the patients, two techniques will be used: standard Polymerase chain reaction amplification with primers flanking the intron 2 fragment of the RFC1 gene and amplification using Repeated Primed Polymerase chain reaction in 3 independent reactions.

DETAILED DESCRIPTION:
A descriptive cross-sectional pilot study that included 50 non-smoking patients between the ages of 30 and 99 years with chronic and / or refractory cough as the only manifestation or associated with gastroesophageal reflux.

All patients will undergo the pertinent studies for the diagnosis of chronic cough, those who meet criteria for suspected gastroesophageal reflux will be asked for an esophageal phmetry and esophageal manometry, according to the usual clinical practice.

Peripheral venous blood sample will be obtained for subsequent genetic analysis.

Vibration sensitivity will be studied in all patients regardless of the presence of mutation.

Those with alterations in vibratory sensitivity or mutations in RFC1 will be referred to the Neurology Service for a complementary neurological evaluation. For the molecular study of the DNA sample of the patients, two techniques will be used: standard Polymerase chain reaction amplification with primers flanking the intron 2 fragment of the RFC1 gene and amplification using Repeated Primed Polymerase chain reaction in 3 independent reactions.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* Aged between 30 and 99 years
* with chronic and / or refractory cough as the only manifestation or associated with gastroesophageal reflux, who have signed the informed consent will be included.

Exclusion Criteria:

* Other causes of cough other than gastroesophageal reflux: pneumological diseases (asthma, Chronic obstructive pulmonary disease, bronchiectasis, tracheomalacia, cystic fibrosis, residual pleural diseases, interstitial diseases, infectious diseases.)
* Upper airway pathologies (rhinitis, sinusitis)
* Foreign bodies
* Smokers or ex-smokers
* Symptoms of associated respiratory allergies
* Severe associated comorbidity.
* Autoimmune disease or systemic inflammatory disease.
* Active immunodeficiency.
* Neoplastic disease.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients, non-smokers, aged between 30 and 99 years, with chronic and / or refractory cough as the only manifestation or associated with gastroesophageal reflux, who have signed the informed consent will be included.
  Chronic cough will be defined as cough lasting more than 8 weeks that is not related to an acute (3 weeks) or subacute (3-8 weeks) process.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Presence of biallelic expansion of AAGGG in RFC1 in patients with chronic cough, regardless of the presence of neurological symptoms | 6 months
  Study of the DNA sample of the patients with two techniques: standard Polymerase chain reaction amplification with primers flanking the intron 2 fragment of the RFC1 gene and amplification using Repeated Primed Polymerase chain reaction in 3 independent reactions.

SECONDARY OUTCOMES:
Phenotypic, functional and inflammatory characteristics of these patients | 12 months
  The tests of the usual clinical practice will be carried out for the study of chronic cough

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Crespo, MD,PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
* Study design (from November 2020 to June 2021): In this phase, the protocol will be elaborated, the study materials will be edited, the database design will be carried out, meetings will be held with the researchers to resolve doubts The logistical aspects will be prepared for the start of the study and the project will be presented to the Hospital's ethics committee.
  * Recruitment period: one year (study start in June 2021): In this phase, patients will be identified, data will be collected and entered. This phase would end in June 2022.
  * Period of analysis of the genetic samples, purification and analysis of the data: this phase is calculated to be carried out in 6 months (June 2022 to December 2022)
  * Period of interpretation of the results and writing of memory: for the publication of the results (December 2023 to June 2024).

REFERENCES:
- [Background] Infante J, Garcia A, Serrano-Cardenas KM, Gonzalez-Aguado R, Gazulla J, de Lucas EM, Berciano J. Cerebellar ataxia, neuropathy, vestibular areflexia syndrome (CANVAS) with chronic cough and preserved muscle stretch reflexes: evidence for selective sparing of afferent Ia fibres. J Neurol. 2018 Jun;265(6):1454-1462. doi: 10.1007/s00415-018-8872-1. Epub 2018 Apr 25. PMID 29696497
- [Background] Szmulewicz DJ, McLean CA, MacDougall HG, Roberts L, Storey E, Halmagyi GM. CANVAS an update: clinical presentation, investigation and management. J Vestib Res. 2014;24(5-6):465-74. doi: 10.3233/VES-140536. PMID 25564090
- [Background] Scriba CK, Beecroft SJ, Clayton JS, Cortese A, Sullivan R, Yau WY, Dominik N, Rodrigues M, Walker E, Dyer Z, Wu TY, Davis MR, Chandler DC, Weisburd B, Houlden H, Reilly MM, Laing NG, Lamont PJ, Roxburgh RH, Ravenscroft G. A novel RFC1 repeat motif (ACAGG) in two Asia-Pacific CANVAS families. Brain. 2020 Oct 1;143(10):2904-2910. doi: 10.1093/brain/awaa263. PMID 33103729
- [Background] Cortese A, Simone R, Sullivan R, Vandrovcova J, Tariq H, Yau WY, Humphrey J, Jaunmuktane Z, Sivakumar P, Polke J, Ilyas M, Tribollet E, Tomaselli PJ, Devigili G, Callegari I, Versino M, Salpietro V, Efthymiou S, Kaski D, Wood NW, Andrade NS, Buglo E, Rebelo A, Rossor AM, Bronstein A, Fratta P, Marques WJ, Zuchner S, Reilly MM, Houlden H. Biallelic expansion of an intronic repeat in RFC1 is a common cause of late-onset ataxia. Nat Genet. 2019 Apr;51(4):649-658. doi: 10.1038/s41588-019-0372-4. Epub 2019 Mar 29. PMID 30926972